CLINICAL TRIAL: NCT03162315
Title: The Value of Progesterone for the Timing of the Embryo Transfer in IVF/ICSI: a Prospective Randomised Trial
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Ghent (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: B670201627451
Record Dates: First submitted 2016-03-23; First posted 2017-05-22 (Actual); Last update posted 2020-04-02 (Actual); Status verified 2019-10

CONDITIONS: Clinical Pregnancy Rate

ARMS (2):
- Fresh embryo transfer (No Intervention): fresh embryo transfer (standard of care)
- Freeze all (Experimental): Vitrification of all embryos and replacement of a thawed embryo in a subsequent cycle
  Interventions: Procedure: Freeze all

INTERVENTIONS:
Procedure: Freeze all
  Arms: Freeze all

SUMMARY:
At the start of the controlled ovarian stimulation as a part of the IVF/ICSI treatment patients are informed about this trial. In case they gave informed consent and they have a progesterone level between 1 and 1.5 ng/ml at the day of the hCG injection, they will be randomised. One group of patients will have a fresh embryo transfer, in the second group all embryos will be cryopreserved and transfered in a subsequent (natural or artificial) cycle. The aim of this study is to compare clinical pregnancy rate between the two groups.

ELIGIBILITY:
Inclusion Criteria:

* IVF/ICSI treatment
* progesterone > 1 ng/ml and ≤ 1.5 ng/ml

Exclusion Criteria:

* > 40 years
* AMH ≤ 1 ng/ml
* Conditions influencing pregnancy rate (e.g. hydrosalphinx, uterus malformation, hyperprolactinemia and other endocrine conditions; with the exception of controlled thyroid function disease)
* no available progesterone value on the day of hCG-injection

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 24 (Actual)
Dates: Start 2016-03; Primary Completion 2018-08-03 (Actual); Study Completion 2018-08-03 (Actual)

PRIMARY OUTCOMES:
Clinical pregnancy rate | 7 gestational weeks

SECONDARY OUTCOMES:
Ongoing pregnancy rate | 25 gestational weeks
Live birth rate | Delivery

CONTACTS AND LOCATIONS:
Overall Officials: Frank Vandekerckhove, MD, PhD, Principal Investigator — University Hospital, Ghent
Locations (1):
- Ghent University Hospital - Department of Reproductive Medicine, Ghent, Belgium

IPD SHARING:
Plan to Share IPD: No